CLINICAL TRIAL: NCT04087512
Title: Comparison of an Instrumented and a Conventional Perturbation-Based Balance Training for Preventing Falls in Older Persons
Brief Title: Instrumented vs. Conventional Perturbation-based Balance Training for Fall Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to sudden Corona pandemic related restrictions and an expiration of funding in case of further delay it was decided to prematurely terminate study recruitment and proceed evaluation with a smaller sample size than intended (n=71 instead n=111).
Sponsor: Leon Brüll (Other)
Collaborators: Humboldt-Universität zu Berlin (Other)
Responsible Party: Sponsor-Investigator, Leon Brüll, M.A., Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AZ Schwe 2019 /1-2
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Fall Risk, Fall Prevention
Keywords: perturbation-based balance training; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors are blinded during baseline-assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instrumented perturbation-based balance training (Experimental)
  Interventions: Other: Training on perturbation treadmill
- Conventional perturbation-based balance training (Experimental)
  Interventions: Other: Exercises of dynamic stability under unstable conditions
- Control (No Intervention)

INTERVENTIONS:
Other: Training on perturbation treadmill — Perturbations into different directions are induced during static and dynamic tasks on a treadmill. Perturbations include announced and unannounced perturbations. Intensity and number of perturbations increases over the course of the intervention based on judgement of participant. Intervention duration: 6 weeks, 3 sessions a week, each session approx. 30 minutes.
  Arms: Instrumented perturbation-based balance training
Other: Exercises of dynamic stability under unstable conditions — The mechanisms of dynamic stability recovery are trained under unstable conditions. Different unstable undergrounds are used to stand on, perform lunges or jumps. Additionally, balance is challenged by different restrictions (e.g. decreased base of support, closed eyes) or therapist-applied perturbations. Intervention duration: 6 weeks, 3 sessions a week, each session approx. 45 minutes.
  Arms: Conventional perturbation-based balance training

SUMMARY:
In the past years, several studies have demonstrated the potential of task-specific perturbation-based balance training (PBT) for preventing falls at age. However, different paradigms of PBT have been investigated so far, while a comparison of these paradigms is lacking. Therefore, in this study, we plan to compare two promising PBT approaches in terms of feasibility and effects on fall risk-associated motor performance: 1. Training of dynamic stability mechanisms in the presence of perturbations induced by unstable surfaces; 2. Technology-supported training on a perturbation treadmill. In addition, both approaches will be compared with a passive control group. One-hundred and eleven participants aged 65 years or older will be randomly assigned to the three arms of the study. As the primary outcome, we will assess fall risk by use of the Brief-BESTest. Secondary outcomes include balance performance, functional performance, force capacity, and more. We hypothesize that both interventions will lead to a significant reduction of fall risk compared to the control group. Additionally, we will explore whether one of the two PBT paradigms is superior regarding feasibility and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Speaks German language
* Home-dwelling or assisted living
* One fall in the past 12 months OR a verified fall risk (based on subjective decreased balance AND extended Short Physical Performance Battery (SPPB) balance testing
* Able to walk at least 20 minutes without aid
* Available for intervention period

Exclusion Criteria:

* Participation in balance training in the previous 3 months
* DemTec ≤ 8 Points
* Body mass index > 30
* Uncorrected vision disorder
* Acute serious neurological disability affecting gait pattern
* Serious sensory disorders
* Severe cardiovascular or metabolic disorders
* Orthopaedic restrictions or diseases
* Strong dizziness
* Current chemotherapy
* Severe respiratory disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Balance performance | Change from baseline to post intervention test (an average of 7 weeks)
  Brief Balance Evaluation Systems Test (Brief-BESTest)

SECONDARY OUTCOMES:
Neuromuscular control during perturbations | Change from baseline to post intervention test (an average of 7 weeks)
  Muscle synergies derived by non-negative matrix factorization from surface electromyography on 13 leg muscles
Reactive balance performance | Change from baseline to post intervention test (an average of 7 weeks)
  Step, stepping, fall-threshold test on Balance Tutor
Static balance performance | Change from baseline to post intervention test (an average of 7 weeks)
  Center of pressure on force plate
Limits of stability | Change from baseline to post intervention test (an average of 7 weeks)
  Limits of stability on force plate
Spatio-temporal gait parameters | Change from baseline to post intervention test (an average of 7 weeks)
  GAITRite System
Functional leg strength (a) | Change from baseline to post intervention test (an average of 7 weeks)
  30 s Chair rise test
Functional leg strength (b) | Change from baseline to post intervention test (an average of 7 weeks)
  Timed Up-and-Go test
Force capacity of knee extensors | Change from baseline to post intervention test (an average of 7 weeks)
  Isometric force test on force plate
Fear of falling | Change from baseline to post intervention test (an average of 7 weeks)
  Short Falls Efficacy Scale-International (Short FES-I); range: 7-28 points, high value indicates high fear of falling
Feasibility of training paradigms | Post intervention test (on average 7 weeks after baseline)
  Acceptance of training questionnaire; range: 1-6 points, high value indicates high acceptance

CONTACTS AND LOCATIONS:
Locations (1):
- Heidelberg University, Network Aging Research, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided